CLINICAL TRIAL: NCT06726694
Title: Assessment of Skeletal, Dental and Soft Tissue Changes in Class II Malocclusion Correction Using the Mini-screw Supported Advanced Molar Distalization Appliance
Brief Title: Class II Malocclusion Correction Using the Mini-screw Supported Advanced Molar Distalization Appliance
Acronym: (AMDA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Distalization
Record Dates: First submitted 2024-12-06; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2020-05

CONDITIONS: Class II Malocclusion
Keywords: Disatlization; class II; growing patient; molar tipping
MeSH Terms: conditions — Overbite

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- class II malocclusion patients (Active Comparator): class II molar relation correction by advanced maxillary molar distalization appliance
  Interventions: Device: class II molar relation correction by advanced molar distalization appliance

INTERVENTIONS:
Device: class II molar relation correction by advanced molar distalization appliance — correction of class II molar relation by a novel miniscrews distalizer
  Other Names: AMDA; miniscrews supported distalizer

SUMMARY:
the primary aim for this clinical trial was to assess the amount of molar distalization

The subjects with the following inclusion criteria:

1. Early permanent dention.
2. Class II division 1 or class II division 2 dental occlusion.
3. Good oral hygiene.
4. No previous orthodontic treatment.
5. No history of serious medical problems such as diabetes or autoimmune disease, allergies or bone disease.
6. Good periodontal support of the upper molar.

DETAILED DESCRIPTION:
Study procedure:

An informed consent was signed by the patients before their enrolment in the current study in which the aim of the study, the methodology and possible complications was clearly described. This research was reviewed by Research Ethics Committee, Faculty of Dentistry, Ain Shams University.

Full orthodontic records were taken for patients who meet the inclusion criteria. These records are:

1. Extra-oral and intra-oral photographs.
2. Orthodontic study cast before after distalization.
3. Panoramic radiograph.
4. Lateral cephalometric radiograph.

Procedure:

1. Bands on first molars are fitted with lingual sheaths.
2. Impression with bands in place is taken and poured into stone model.
3. Positioning the appliance on the model by inserting the palatal extension in the lingual sheaths of the molar bands, where the arch wire should be apical and parallel to the occlusal plane. The width of the horseshoe type palatal arch wire is adjusted to fit palatal width.
4. The mesial stop screws are moved distally to fully compressed the coil spring encased in the tubing system and the distal stop screws are screwed in place to stabilize the tubing system on the archwire.
5. The final length of the palatal archwire is determined by marking its distal end with a pencil, leaving approximately 8-10mm extended out of the distal screw.
6. Remove the appliance and cut off the distal end at the mark and bend or loop is formed on each distal end to act as mechanical stop to prevent any distalization beyond this point and to avoid any tissue irritation. Alternatively, or in addition, a small amount of light cured resin can be added to the end to ensure that the molar cannot slip out of the wire.
7. The appliance is disinfected and inserted into the patient mouth, ensuring that it parallel to the occlusal plane and the two symmetrical loops are posterior to the incisive foramen.
8. The wire extensions welded on the tubing system are inserted into the lingual sheath of the molar band and secured in position with SS ligature wire.
9. The palatal is rinsed with a 0.02% chlorohexidine solution.
10. Small amount of local anaesthesia is applied to the soft tissue of the palatal.
11. 2 miniscrews implants are inserted through the two symmetrical closed loops of the horseshoe type palatal arch wire using especial screwdriver at the paramedian region of the palate.
12. A small portion of light-cure resin can be added to cover the top of each implant head plus the ending of the ligature wires and the loops of the palatal arch wire to avoid plaque accumulation.
13. Activation of the AMDA by unscrewing the distal screws to allow free distal sliding of the posterior part of the tubing system, the mesial stop screws are not altered.
14. Following initial activation of the AMDA, the patient is monitored at 4-week intervals and reactivation is done when force decreases until Class I molar relationship is obtained

Adverse event reporting:

• acceptable discomfort and mild to moderate pain.

Methods of assessment:

1. The rate of tooth movement was analyzed using computer software on digital models obtained by scanning orthodontic study casts taken before and after molar distalization. When a Class I molar relationship is obtained distalization will be considered complete, this was assessed visually.
2. Lateral cephalometric radiograph was obtained before and after molar distalization for all participants.
3. All data was tabulated and statistically analyzed.

ELIGIBILITY:
The subjects were selected to fulfil the following inclusion criteria:

1. Early permanent dention.
2. Class II division 1 or class II division 2 dental occlusion.
3. Good oral hygiene.
4. No previous orthodontic treatment.
5. No history of serious medical problems such as diabetes or autoimmune disease, allergies or bone disease.
6. Good periodontal support of the upper molar.

Exclusion criteria:

1. Patients with severe crowding requiring extraction.
2. Vertical growth patterns.
3. Syndromic patients.
4. Vulnerable groups.

Ages: 11 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
amount of molar distalization | 8 months
  measuring the amount of molar distalization in millimeter by cephalometric analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Abbasia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
inclusion criteria study procedures conclusions
Supporting Information: Study Protocol, ICF
Time Frame: 1| 2| 2025
  1| 5 | 2025
Access Criteria: Noha Ibrahim google drive 5 | 2025

REFERENCES:
- [Background] Papadopoulos MA. Efficient Distalization of Maxillary Molars with Temporary Anchorage Devices for the Treatment of Class II Malocclusion. Turk J Orthod. 2020 Aug 20;33(3):197-201. doi: 10.5152/TurkJOrthod.2020.20064. eCollection 2020 Sep. PMID 32974067